CLINICAL TRIAL: NCT04468139
Title: The Study of Quadruple Therapy Zinc, Quercetin, Bromelain and Vitamin C on the Clinical Outcomes of Patients Infected With COVID-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Amr kamel khalil Ahmed, director of mobile team tuberculosis ghubera, tuberculosis control program, Ministry of Health, Saudi Arabia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-95M
Record Dates: First submitted 2020-07-05; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Quercetin; Bromelains; Zinc; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Quercetin (Experimental): Quercetin 500 g of quercetin Quercetin will be administered orally once daily, in the morning before breakfast for 5-10 days or patient improves or discharged
  Interventions: Drug: Quercetin; Dietary Supplement: bromelain; Drug: Zinc; Drug: Vitamin C

INTERVENTIONS:
Drug: Quercetin — Dietary Supplement: Quercetin Treatment a daily dose of quercetin (500 mg) will be taken orally by proven COVID-19 cases intervention
Dietary Supplement: bromelain — Dietary Supplement:Bromealin Treatment a daily dose of bromelain(500 mg) will be taken orally by proven COVID-19 cases intervention
Drug: Zinc — zinc 50 mg orally daily dose will be taken orally by proven COVID-19 cases intervention
Drug: Vitamin C — vitamin c 1000 mg orally daily by proven COVID-19 cases intervention

SUMMARY:
There are currently no antiviral drugs with proven efficacy nor are there vaccines for its prevention. Unfortunately, the scientific community has little knowledge of the molecular details of SARS-CoV-2 infection. The drugs we are chosen are used as clinical trials for antiviral and there is no proven guide for specificity and effectiveness against the virus so the results are different Now the clinical trials and research authorities are work speedily to target the most proven treatment for the virus so anything is infantile until now. the covid-19 with time be more explained by scientists it is steroid response disease and cause thromosis and cytokine storm , the aim of the study to inhibit viral replication and decrease the severity of the disease as antiviral and anticytokine storm , antithrombosis Zinc is a mineral element needed to regulate adaptive immune cells' functions. Higher level of intracellular zinc showed to increase intracellular pH; which affect on RNA-dependent RNA polymerase and decrease replication mechanism of RNA viruses. Therefore, drugs that described as zinc ionophores could be used with zinc supplement to act as antiviral against many RNA viruses including SARS-CoV-2 Quercetin is natural compound act as zinc ionophore to cause zinc influx intracellular.

Quercetin is a safe natural anti-oxidant and anti-inflammatory polyphenolic compound that found in various natural sources include onion, red grapes, honey and citrus fruits. It was shown that quercetin has the ability to chelate zinc ions and act as zinc ionophore. Therefore, quercetin could have antiviral activity against many RNA viruses . Quercetin, a flavonoid found in fruits and vegetables, has unique biological properties that may improve mental/physical performance and reduce infection risk ; These properties form the basis for potential benefits to overall health and disease resistance, including anti-carcinogenic, anti-inflammatory, antiviral, antioxidant, and psychostimulant activities, as well as the ability to inhibit lipid peroxidation, platelet aggregation and capillary permeability, and to stimulate mitochondrial biogenesis .There are various studies that report the immunomodulatory effect of bromelain . Bromelain activates natural killer cells and augments the production of granulocyte-macrophage-colony stimulating factor, IL-2, IL-6 and decreases the activation of Thelper cells. Thus, bromelain decreases the majority of inflammatory mediators and has demonstrated a significant role as an anti-inflammatory agent in various conditions Vitamin C is known as an essential anti-oxidant.,and enzymatic co-factor for physiological reactions such as hormone production, collagen synthesis and immune potentiation . Naturally, an insufficiency of vitamin C leads to severe injuries to multiple organs, especially to the heart and brain, since they are both highly aerobic organs that produce more oxygen radicals. In fact, studies of in vivo effect on vitamin C are difficult since most animals, except human and some primate, are capable of synthesizing vitamin C endogenously

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. positive confirmed PCR covid-19
3. moderate to severe cases
4. obtained consent
5. must be able to swallow tablets

Exclusion Criteria:

1. Patients who live outside Saudia Arabia
2. Pregnant women: Current known pregnancy positive pregnancy test.
3. Lactating women.
4. Documented allergy to pineapple or to quercetin
5. Documented history of mental illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2020-07-20 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
days of stay at hospital after treatment and discharge | 28 days
  speed the days of recovery and discharge from hospital
serum zinc before and after treatment | 5-10 days
  the level of serum zinc is very important especially at chronic diseases

SECONDARY OUTCOMES:
questionnaire including parameters like BMI,,smoking , underling diseases, immunological treatment , | 28 days
  according to questionnaire including BMI, smoking , underlying diseases like hypertension, diabetes , asthmatic , ..etc
day of negative conversion for nasopharyngeal swab for rt-PCR FOR covid-19 | 28 days
  day of negative conversion for nasopharyngeal swab for rt-PCR FOR covid-19

CONTACTS AND LOCATIONS:
Overall Officials: Hiba Hamadelnil elsaeed, Study Director — Netherlands: Ministry of Health, Welfare and Sports
Locations (1):
- Ministry of health.First health cluster ,Riaydh, Riyadh, Saudi Arabia